CLINICAL TRIAL: NCT00079768
Title: Effects of a T Cell-Depleting Monoclonal Antibody, Alemtuzumab, in Patients With Inclusion Body Myositis: A Pilot Clinicopathological Study
Brief Title: Alemtuzumab to Treat Sporadic Inclusion Body Myositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Marinos C. Dalakas, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040133; 04-N-0133
Record Dates: First submitted 2004-03-12; First posted 2004-03-12 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2009-01

CONDITIONS: Myositis, Inclusion Body
Keywords: Inflammation; Myositis; Humanized Monoclonal Antibody; Cytotoxic T Cells; Endomysial T Cells; Alemtuzumab; Monoclonal Antibodies; IBM; Anti-CD 52; Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body; Inflammation; Myositis | interventions — Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab (Campath)

SUMMARY:
This study will examine the safety and effectiveness of alemtuzumab (Campath® (Registered Trademark)) for improving muscle strength in patients with sporadic inclusion body myositis (s-IBM). The most common inflammatory muscle disease in people over the age of 50, s-IBM progresses steadily, leading to severe weakness and wasting of the muscles in the arms and legs. The cause of s-IBM is not known, but it may be an autoimmune disease, in which the body's immune cells (white blood cells) attack and destroy parts of muscle. Alemtuzumab is a laboratory-made antibody currently approved to treat certain leukemias. It has also been used to treat patients with autoimmune conditions such as rheumatoid arthritis, vasculitis, multiple sclerosis, and tissue rejection associated with transplantation. Alemtuzumab destroys white blood cells that have a protein called CD52 on their surface and that might be among the cells attacking muscle.

Patients with s-IBM are eligible for this study. Candidates are screened with physical and neurological examinations, blood tests, and an electrocardiogram. Participants undergo the following tests and procedures:

* Campath administration: Patients are admitted to the NIH Clinical Center for 1 to 1-1/2 weeks for intravenous infusions of Campath, given every other day for a total of 4 infusions.
* Follow-up visits after infusions: Patients are monitored for up to 1 year with periodic blood tests, physical and neurological examinations, medical history, muscle strength measurements, and a review of symptoms, including the ability to perform daily living activities.
* Lymphapheresis: Patients undergo this procedure for collecting large numbers of white blood cells twice - once at the beginning of the study and again after 6 months. Blood is removed through a needle in an arm vein and flows through a machine that separates it into its components by centrifugation (spinning). The white cells and plasma are removed and the red cells and platelets are returned to the patients through the same needle or through another needle in the other arm.
* Muscle biopsy: Muscle biopsies are done in the operating room under local anesthetic. A small incision is made in the thigh or upper arm and a small piece of muscle is removed. Biopsies are done at the beginning of the study and again after 6 months.

DETAILED DESCRIPTION:
Sporadic Inclusion-Body Myositis (s-IBM) is the most common muscle disease in patients above the age of 50 years. It is an inflammatory myopathy mediated by sensitized, cytotoxic CD8+ T cells that clonally expand in situ and invade MHC-I-expressing muscle fibers. The antigen recognized by the T cells is unknown. The disease is progressive, resists the currently available immunotherapies and leads to wheelchair confinement. Applying therapeutic strategies with agents that deplete T cells clones and investigating the antigenic specificity of the endomysial T cells is expected to enhance our understanding of the cause of s-IBM and lead to clinical improvement. The present study is designed to: a) test in a pilot study the safety, T cell depletion of the endomysial T cells and clinical efficacy of the monoclonal antibody Alemtuzumab in 20 patients with s-IBM followed for 12 months by serial quantitative assessment of muscle strength; b) explore the spectrum of the antigens recognized by the T cells extracted from the muscle biopsy specimens by searching for immune dominant peptides using positional scanning synthetic combinational peptide libraries, before and after therapy; and c) determine the reciprocal relationship between clinical response and endomysial inflammatory mediators before and after treatment. It is anticipated that the study may lead to identification of putative antigens that trigger the disease, clarify the significance of the inflammation and amyloid deposits in muscle fiber injury and provide a novel therapy for s-IBM patients.

ELIGIBILITY:
* Only patients who are currently enrolled in protocol 02-N-0121 Study of Immune Dysregulation in Patients with Sporadic Inclusion Body Myositis (s-IBM) will be considered for enrollment in protocol 04-N-0133.

INCLUSION CRITERIA:

Patients with confirmed diagnosis of s-IBM willing to undergo therapy with Alemtuzumab.

Willingness and legal ability to give and sign informed study consent.

Willingness to travel to the Clinical Center for planned studies and treatment as required by protocol.

Men and women of reproductive potential must agree to use an acceptable method of birth control during and for six months after completion of treatment.

Availability of tissue for testing. This will include muscle and peripheral blood lymphocytes isolated through routine lymphocytapheresis or phlebotomy.

EXCLUSION CRITERIA:

Immunosuppressive drug therapy at the time of or 6 months prior to enrollment. Specifically, candidates may not be taking Prednisone, cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, anti-lymphocyte agents, cyclophosphamide methotrexate, or other agents whose concomitant use may enhance the toxicity of Alemtuzumab.

Any medical or personal difficulties that precludes serial follow-up visits.

Any active malignancy.

Significant coagulopathy or requirement for anticoagulation therapy that would contraindicate protocol.

Platelet count less than 100,000/mm(3).

Hemoglobin less than 9.0 mg/dl.

Any known immunodeficiency syndrome included HIV infection.

Any history of cardiac insufficiency, major vascular disease, or unstable coronary artery disease.

Any history of systemic or pulmonary edema.

Any history of previous treatment with monoclonal antibodies or sensitivity to the study drug (Alemtuzumab), pre-medication regimen, or prophylactic agents.

History of chronic hypotension (SBP less than 100 mmHg).

Any medical condition that would likely increase the risk of side effects of the study drug or confound the interpretation of the data including active infections.

Pregnancy and active nursing (breast feeding).

History of uncontrolled thyroid disease or a history of autoimmune thyroiditis.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change in the muscle strength at 6 months by 15%.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dalakas MC. Polymyositis, dermatomyositis and inclusion-body myositis. N Engl J Med. 1991 Nov 21;325(21):1487-98. doi: 10.1056/NEJM199111213252107. No abstract available. PMID 1658649
- [Background] Dalakas MC, Sonies B, Dambrosia J, Sekul E, Cupler E, Sivakumar K. Treatment of inclusion-body myositis with IVIg: a double-blind, placebo-controlled study. Neurology. 1997 Mar;48(3):712-6. doi: 10.1212/wnl.48.3.712. PMID 9065553
- [Background] Dalakas MC, Koffman B, Fujii M, Spector S, Sivakumar K, Cupler E. A controlled study of intravenous immunoglobulin combined with prednisone in the treatment of IBM. Neurology. 2001 Feb 13;56(3):323-7. doi: 10.1212/wnl.56.3.323. PMID 11171896
- [Derived] Dalakas MC, Rakocevic G, Schmidt J, Salajegheh M, McElroy B, Harris-Love MO, Shrader JA, Levy EW, Dambrosia J, Kampen RL, Bruno DA, Kirk AD. Effect of Alemtuzumab (CAMPATH 1-H) in patients with inclusion-body myositis. Brain. 2009 Jun;132(Pt 6):1536-44. doi: 10.1093/brain/awp104. Epub 2009 May 19. PMID 19454532